CLINICAL TRIAL: NCT05973292
Title: Endocrowns in Anterior Teeth: Effect of Cementation Protocols and Restorative Materials on the Clinical Performance of the Restorations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Nehal Samra, Assistant Lecturer- Prosthodontic Department- Faculty of Dentistry, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M01160321
Record Dates: First submitted 2023-07-26; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Endodontically Treated Teeth; Anterior Teeth
Keywords: Digital Dentistry, E-max, MDP, Zirconia
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Intervention Model Description: All patients received their treatment at the same time. Follow-up periods were parallel for all participants.
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcome assessors and participants were blinded throughout the whole procedure. The dentist practitioner was responsible for all clinical procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group ZA (Experimental): Participants received Zirconia anterior endocrowns. Endocrowns were cemented with MDP-containing primer+ MDP-containing resin cement.
  Interventions: Other: resin cement containing phosphate ester monomer 10-methacryloyloxydecyl dihydrogen phosphate
- Ggroup ZB (Experimental): Participants received Zirconia anterior endocrowns. Endocrowns were cemented with MDP-containing primer+ Non-MDP-containing resin cement.
  Interventions: Other: Non MDP containg resin cement
- Group EA (Experimental): Participants received E-max anterior endocrowns. Endocrowns were cemented with MDP-containing primer+ MDP-containing resin cement.
  Interventions: Other: resin cement containing phosphate ester monomer 10-methacryloyloxydecyl dihydrogen phosphate
- Group EB (Experimental): Participants received E-max anterior endocrowns. Endocrowns were cemented with MDP-containing primer+ Non-MDP-containing resin cement.
  Interventions: Other: Non MDP containg resin cement

INTERVENTIONS:
Other: resin cement containing phosphate ester monomer 10-methacryloyloxydecyl dihydrogen phosphate — Adhesive resin cement containing an MDP agent that is added to bonding agents to enhance bonding to ceramics like Ziconia and E-max
  Other Names: Panavia SA
  Arms: Group EA; Group ZA
Other: Non MDP containg resin cement — Adhesive resin cement not containing an MDP agent
  Other Names: Duo-link Universal
  Arms: Ggroup ZB; Group EB

SUMMARY:
Rehabilitation of anterior endodontically treated teeth with significant coronal damage has been problematic. Adopting endocrown design to treat teeth with this condition is still under investigation. To address this issue, the USPHS criteria were adopted to assess the anterior endocrown restorations manufactured using various ceramic materials and cemented with different protocols.

DETAILED DESCRIPTION:
40 participants with anterior endodontically treated maxillary central incisors were enrolled to restore their teeth with esthetic restorations Patients were divided into two groups, zirconia and e-max groups. Each group was, further subdivided into two groups following the cementation protocol. Patients were evaluated immediately (baseline) and at. The clinical marginal accuracy measurements were carried out for all groups at baseline, 3, 6, 9, 12, and 18 months and evaluated by 3 investigators using Modified (USPHS). The patients' satisfaction and potential postoperative discomfort were also assessed and recorded during the same periods. All qualitative data were displayed as frequency (N) and Percentages (%). The chi-square test was utilized for qualitative data comparisons.

Results:

As to marginal integrity and patient satisfaction, no significant difference were revealed regarding all scores at different intervals as P>0.05.

Conclusions:

According to the findings of this study, ceramic endocrowns offer a promising restorative solution for the rehabilitation of anterior endodontically treated teeth. Additionally, regardless of the presence of the MDP monomer in its composition, using adhesive resin cement achieved highly successful results when used with MDP-based ceramic primers.

ELIGIBILITY:
Inclusion Criteria:

* • Freshly extracted teeth.

  * Completely formed apices
  * Minimum root length of 14mm (± 0.5) measured from the cement-enamel junction to the root apex.
  * Straight roots.
  * Teeth with single root canal.
  * Sound teeth with no cracks or fractured parts in its crown or root.
  * Absence of any carious lesions.
  * No signs of internal or external root resorption.
  * Similar bucco-lingual (BL) and mesio-distal (MD) dimensions as determined with a digital caliper.

Exclusion Criteria:

* • Previously endodontically treated teeth.

  * Markedly curved roots.
  * Root contains more than one canal.
  * Presence of canal calcifications or pulp stones.
  * Internal or external root resorption.
  * Presence of cracks, fractures or caries.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Marginal Integrity | 3-6-9-12 Months
  Using a dental mirror and a dental explorer, endocrowns were checked from every aspect, buccal, mesial, distal and lingual to detect any marginal discontinuity, fractures, or gaps. Endocrown evaluation was carried out against The Modified USPHS criteria

SECONDARY OUTCOMES:
Patient Satisfaction | 3-6-9-12 Months
  Each patient was asked about his opinion regarding the restoration. Patients' answers and/or complaints were assessed and recorded against the USPHS criteria

CONTACTS AND LOCATIONS:
Overall Officials: Lamia Dawood, Professor, Study Director — Professor of Fixed Prosthodontics, Faculty of Dentistry, Mansoura University, Mansoura, Egypt.
Locations (1):
- Faculty of Dentistry,Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt